CLINICAL TRIAL: NCT01007149
Title: A 16-week Treatment, Multicenter, Randomized, Double Blind, Placebo-controlled, Parallel-group Study to Assess the Effect of Omalizumab on the Expression of FcεRI Receptors of Blood Basophils and Dendritic Cells in Patients With Severe Persistent Non-atopic Asthma, Uncontrolled Despite Optimal Therapy
Brief Title: Effect of Omalizumab in Patients With Severe Persistent Non-atopic Uncontrolled Asthma
Acronym: NATAIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CIGE025AFR05; 2009-010937-38 (EudraCT Number)
Record Dates: First submitted 2009-10-30; First posted 2009-11-03 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Severe asthma,; non-atopic,; omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Omalizumab (Experimental): Participants received subcutaneous injections of omalizumab every 2 weeks or every 4 weeks; dosage dependent on IgE level and body weight.
  Interventions: Drug: omalizumab
- Placebo (Placebo Comparator): Participants received subcutaneous injections of placebo to omalizumab every 2 weeks or every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: omalizumab — Omalizumab was supplied in 5mL vials with solution for subcutaneous injection.
  Arms: Omalizumab
Drug: Placebo — Placebo was supplied in vials with solution for subcutaneous injection.
  Arms: Placebo

SUMMARY:
This study will assess the change in the expression of FcεRI receptors of blood basophils and dendritic cells after 16 weeks of treatment with omalizumab as compared with placebo, in adult patients with non-atopic severe persistent asthma, uncontrolled despite optimal therapy.

ELIGIBILITY:
Inclusion Criteria:

Severe persistent asthma with the following characteristics:

* Uncontrolled according to Global Initiative for Asthma (GINA) 2007 guidelines and at least 2 exacerbations having required systemic corticosteroid and/or at least 1 hospitalization or emergency room visit in the past year.
* Treated with high-dose inhaled corticosteroid (i.e. > 1,000 µg beclometasone dipropionate equivalent per day) plus inhaled long-acting β2 agonist (with or without maintenance oral corticosteroid).
* Non-atopic, i.e. negative blood multiallergic testing and negative Aspergillus-specific IgE-radio allergosorbent blood test and negative skin prick tests to a battery of common aeroallergens

Exclusion Criteria:

* Current smokers or smoking history stopped for less than 3 years or > 10 pack years.
* Asthma exacerbation during the 4 weeks prior to randomization.
* Active lung disease other than non-atopic asthma.
* Patients with an active cancer, a suspicion of cancer or any history of cancer with less than 5 disease free years.
* Pregnant or nursing (lactating) women.
* Treatment with omalizumab.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- France (10):
  - Novartis Investigative Site, Arnaud de Villeneuve
  - Novartis Investigative Site, Béthune
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clamart
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Suresnes
  - Novartis Investigative Site, Toulouse

REFERENCES:
- [Derived] Garcia G, Magnan A, Chiron R, Contin-Bordes C, Berger P, Taille C, Devouassoux G, de Blay F, Couderc LJ, Didier A, O'Callaghan DS, Girodet PO, Bourdeix I, Le Gros V, Humbert M. A proof-of-concept, randomized, controlled trial of omalizumab in patients with severe, difficult-to-control, nonatopic asthma. Chest. 2013 Aug;144(2):411-419. doi: 10.1378/chest.12-1961. PMID 23579324

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 patients were screened. 41 patients received study medication.
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 20 | 21
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Administrative problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.67) | 54.6 (12.78) | 54.8 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Expression of FcεRI Receptors of Blood Basophils
Description: Venous blood samples were collected at screening and at Week 16. Flow cytometry analysis determined the FcεRI receptors expression of blood basophils (mean fluorescence intensity(MFI)). Relative change in mean fluorescence intensity at the end of study was expressed as a percentage of baseline value.
Time Frame: Baseline and 16 weeks
Population: Intent to Treat FcεRI analyzable population - all randomized patients who received at least one dose of study drug and had at least one post-baseline efficacy assessment, and who had a valid baseline and post-treatment measurement of FcεRI
Measure: Mean (Standard Deviation); unit: Percent change in MFI
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Percent change in MFI | -84.4 (17.80) | 27.7 (87.90)

2. Secondary Outcome: Change in Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO was measured at baseline, and after 4, 8, 12 and 16 weeks of treatment. Absolute change in FeNO was expressed at each time point versus baseline value.
Time Frame: Baseline and 4, 8, 12 and 16 weeks
Population: Intent to Treat population - all randomized patients who received at least one dose of study drug and had at least one post-baseline efficacy assessment. During different time points, participants with observations at that time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 19 | 20
parts per billion (ppb)
  Week 4 (N = 19, 19) | 2.5 (21.28) | -5.9 (29.72)
  Week 8 (N = 18, 20) | 4.3 (25.48) | -7.4 (30.19)
  Week 12 (N = 19, 18) | 1.0 (17.29) | 1.3 (30.26)
  Week 16 (N = 18, 19) | 2.4 (18.19) | 0.7 (17.57)

3. Secondary Outcome: Change From Baseline in Induced Sputum Eosinophil Count
Description: The induced sputum eosinophil count was measured in a subset of patients in selected centers. Sputum samples were collected at screening and Week 16. Sputum eosinophil count was expressed as a percentage of total nonsquamous cells. Absolute change in sputum eosinophil count was expressed versus baseline value.
Time Frame: Baseline and 16 weeks
Population: Intent to Treat population - all randomized patients who received at least one dose of study drug and had at least one post-baseline efficacy assessment. Only patients with measurements at both baseline and week 16 were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage of total nonsquamous cells
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 9 | 6
Percentage of total nonsquamous cells | -10.2 (32.38) | 2.2 (10.94)

4. Secondary Outcome: Change From Baseline in Score of the Shortened Version of the Asthma Control Questionnaire (Symptoms Plus Short-acting β2-agonist)
Description: The shortened version of the asthma control questionnaire (symptoms plus β2-agonist) consists of 6 subscores (nighttime waking, symptoms on waking, activity limitation, shortness of breath, wheeze and rescue short-acting β2-agonist use) between 0 and 6 (0 = no impairment; 6 = maximum impairment) and a total score between 0 and 6 (subscores mean value). Absolute change in total score and subscores count was expressed versus baseline value. A decrease in score indicates improvement.
Time Frame: Baseline and 16 weeks
Population: Intent to Treat Population - all randomized patients who received at least one dose of study drug and had at least one post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Score units
  Total score | -0.5 (0.98) | -0.5 (1.43)
  Nighttime waking | 0.1 (1.61) | -0.8 (1.69)
  Symptoms on waking | -0.6 (1.32) | -0.9 (1.73)
  Activity limitation | -0.7 (1.34) | -0.5 (1.94)
  Shortness of breath | -0.9 (1.29) | -0.6 (1.75)
  Wheeze (N = 19, 21) | -0.8 (1.62) | -0.3 (1.79)
  Use of rescue short-acting β2-agonist | -0.3 (0.57) | 0.3 (1.45)

5. Secondary Outcome: Change From Baseline in Nasal Symptom Global Score and Individual Components
Description: Nasal symptom score calculated from six scales assessing the nasal symptom severity (sneezing, runny nose, congestion, itchy nose, postnasal drip and nasal symptoms overall). These six scores were rated on a scale from 1 to 7, with 7 being the worst rating. Absolute changes in these six scores were expressed versus baseline values. A negative change indicates improvement. The range of the global score was from 1 to 7, since this is the mean value of all the subscores.
Time Frame: Baseline and 16 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Score units
  Global score | -0.8 (0.74) | -0.3 (1.38)
  Sneezing | -1.1 (1.10) | -0.4 (1.12)
  Runny nose | -0.9 (1.20) | -0.6 (1.83)
  Congestion | -0.6 (1.39) | -0.7 (2.24)
  Itchy nose | -0.4 (0.84) | 0.1 (1.92)
  Postnasal drip | -0.6 (1.50) | 0.3 (1.37)
  Nasal symptoms overall | -1.2 (1.44) | -0.2 (1.81)

6. Secondary Outcome: Physician and Patient Global Evaluation of Treatment Effectiveness
Description: The GETE is an assessment of asthma symptoms controlled in response to asthma treatment. The evaluation was performed independently by both investigator and patient using the same 5 point scale. The scale points are: excellent, good, moderate, poor and worsening. A good or excellent response is suggested as a means of defining a patient who has responded to treatment.
Time Frame: 16 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Participants
  Physician's evaluation - Excellent | 2 | 1
  Physician's evaluation - Good | 6 | 4
  Physician's evaluation - Moderate | 3 | 8
  Physician's evaluation - Poor | 9 | 6
  Physician's evaluation - Worsening | 0 | 2
  Patient's evaluation - Excellent | 2 | 0
  Patient's evaluation - Good | 7 | 5
  Patient's evaluation - Moderate | 6 | 9
  Patient's evaluation - Poor | 5 | 4
  Patient's evaluation - Worsening | 0 | 2

7. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline to 16 Weeks
Description: Spirometry was conducted according to internationally accepted standards. At least three maneuvers were performed at each sampling timepoint. The FEV1 recorded was taken from the maneuver obtained from the single best test curve. The best test curve was defined as the spirogram that gave the largest FEV1.
Time Frame: Baseline and 16 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Liters | 0.25 (0.38) | 0.00 (0.20)

8. Secondary Outcome: Number of Patients With at Least One Asthma-related Event Over 16 Weeks
Description: Asthma-related events were: unscheduled medical visits, emergency room visits and hospitalizations. Details of exacerbations requiring oral or IV corticosteroids were recorded at each visit.
Time Frame: 16 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 21
Participants | 9 | 11

9. Primary Outcome: Change From Baseline in the Expression of FcεRI Receptors of Dendritic Cells
Description: Venous blood samples were collected at screening and at Week 16. Flow cytometry analysis determined the FcεRI receptors expression of dendritic cells (mean fluorescence intensity (MFI)). Relative change in mean fluorescence intensity at the end of study was expressed as a percentage of baseline value.
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change in MFI
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 19 | 20
Percent change in MFI | -56.7 (19.74) | 24.8 (111.71)

ADVERSE EVENTS:
Description: Safety population - all patients who received at least one dose of study drug and had at least one post-baseline safety assessment
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/21
Other Adverse Events (participants affected / at risk) | 16/20 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=20) | Placebo (N=21)
Myocardial infarction (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=20) | Placebo (N=21)
Tachycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Face oedema (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Ear infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Paraesthesia (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.